CLINICAL TRIAL: NCT03608644
Title: Predictive Factors of Outcome of Mechanical Thrombectomy After Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelhady Hamed Mohamed, Principal Investigator, Assiut University
Other Study IDs: PFOOOMTAAIS
Record Dates: First submitted 2018-07-09; First posted 2018-08-01 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Predictive factors of outcome of mechanical thrombectomy after acute ischemic stroke

DETAILED DESCRIPTION:
Acute ischemic stroke is one of the most common causes of disability, dementia and death in developing world. In Egypt, the total lifetime prevalence of ischemic stroke was 7.2/1,000 in the population aged 20 years and more . Although the intravenous thrombolysis is a treatment option within ≤ 4.5 hours after stroke onset, the mechanical thrombectomy can be performed within a more extended time window. A positive results of 5 recent randomized clinical trials are driven mainly from patients treated by mechanical thrombectomy within 6 hours from onset and they demonstrated a clear benefit for mechanical thrombectomy in combination with intravenous thrombolysis. More recent two randomized clinical trials DAWN and DEFUSE 3 demonstrated an overall benefit in functional outcome at 90 days in patients treated with mechanical thrombectomy within 6 to 24 hours or 6 to 16 hours form onset respectively with special criteria. A major issue remains as to identifying patients which likely to benefit from mechanical thrombectomy to improve selection and subsequently clinical prognosis .

These factors include:-

1. Time of presentation.
2. Age.
3. Clinical presentation.
4. Risk factors include Hyperglycemia, peripheral vessel disease, atrial fibrillation, coronary heart disease, hyperlipidemia, smoking, and history of pervious stroke,
5. Socioeconomic status.
6. Collateral and stroke core. In this study the investigators will evaluate prognostic factors influencing angiographic and clinical outcomes at discharge and at three months after mechanical thrombectomy of acute ischemic stroke within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Cerebral infarction in the anterior or posterior circulation (intracranial internal carotid artery, M1 or M2 middle cerebral artery, basilar or vertebral arteries) proven by Computed tomography angiography
3. With or without intravenous thrombolysis
4. Access to endovascular treatment within 24 hours from onset.
5. In selected patients with acute ischemic stroke within 6 to 24 hours of onset must meet DAWN or DEFUSE 3 eligibility criteria.

Exclusion Criteria:

1. Proven occlusion of the cervical carotid artery
2. Disability prior to the stroke (modified ranking scale >3)
3. Opposition of the patient or their family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute ischemic stroke
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
The outcomes of mechanical thrombectomy after acute ischemic stroke within three months | 3 months
  Modified Rankin Scale (mRS) for measuring the degree of disability